CLINICAL TRIAL: NCT00380900
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Test Article or Placebo Administered Orally to Healthy and Osteoarthritis Subjects.
Brief Title: Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses in Healthy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 3189A1-102
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Healthy Subjects; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Drug: AGG-523

SUMMARY:
The purpose of this study is to evaluate the safety and tolerbility of ascending multiple oral doses of AGG-523 in healthy subjects and in subjects with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women, aged 18 to 40 years and subjects with osteoarthritis of the knee, aged 40 to 75 years.
* Women must be of non-childbearing potential, defined as surgically sterile with documentation of ultrasound.
* Must be nonsmoker or smoke less than 10 cigarettes per day.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-07; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Assess the safety of multiple doses of AGG-523 administered to subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Philadelphia, Pennsylvania, United States